CLINICAL TRIAL: NCT02335203
Title: The Effect of Neoadjuvant Depot Medroxyprogesterone Acetate on Glandular Cellularity in Women With Complex Atypical Hyperplasia or Grade 1-2 Endometrial Adenocarcinoma Awaiting Hysterectomy
Brief Title: The Effect of Neoadjuvant DMPA on Glandular Cellularity in Women Awaiting Hysterectomy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Women and Infants Hospital of Rhode Island (Other)
Responsible Party: Principal Investigator, Stephen Fiascone, M.D., MD in Department of Medical Education; OB/GYN Residency Program, Women and Infants Hospital of Rhode Island
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 14-0099
Record Dates: First submitted 2014-12-22; First posted 2015-01-09 (Estimated); Last update posted 2016-09-20 (Estimated); Status verified 2016-09

CONDITIONS: Grade 1 Endometrial Endometrioid Adenocarcinoma; Grade 2 Endometrial Endometrioid Adenocarcinoma; Complex Atypical Endometrial Hyperplasia
MeSH Terms: interventions — Medroxyprogesterone Acetate; N,N-dimethyl-4-anisidine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Depot medroxyprogesterone acetate (Experimental): Women randomized to receive one intramuscular injection of 400mg depot medroxyprogesterone acetate prior to hysterectomy.
  Interventions: Drug: Depot medroxyprogesterone acetate
- Placebo injection (Placebo Comparator): Women randomized to receive one intramuscular injection of 1mL normal saline prior to hysterectomy.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Depot medroxyprogesterone acetate — One injection intragluteally of 400mg depot medroxyprogesterone acetate at the time of the patient's first visit with the Program in Womens' Oncology
  Other Names: Depo Provera; DMPA
  Arms: Depot medroxyprogesterone acetate
Other: Placebo — One injection intragluteally of 1mL Normal Saline (0.9% Sodium Chloride) at the time of the patient's first visit with the Program in Womens' Oncology
  Other Names: 0.9% Sodium Chloride
  Arms: Placebo injection

SUMMARY:
Objective: To compare pre- and post-treatment glandular cellularity in women with complex atypical hyperplasia or grade 1-2 endometrial adenocarcinoma who are treated with intramuscular depot medroxyprogesterone acetate (DMPA) versus placebo injection prior to hysterectomy. The secondary objective is to compare various other outcomes including molecular, histologic, pathologic and clinical endpoints in women treated with DMPA versus placebo prior to hysterectomy.

Hypothesis: Patients treated with DMPA will have significantly decreased glandular cellularity post-treatment when compared to patients treated with placebo injection. Patients treated with DMPA will exhibit previously described changes in molecular tumor marker expression patterns and other characteristic histologic changes. Patients treated with DMPA will report less bothersome vaginal bleeding prior to surgery when compared to patients treated with placebo injection.

Study Design: Double blinded randomized controlled trial

Population: Women being treated at the Women and Infants Program in Women's Oncology who have a biopsy-proven diagnosis of complex atypical hyperplasia or grade 1-2 endometrial adenocarcinoma with disease clinically confined to the uterus, with a plan to undergo hysterectomy.

Study Period: February 2015 to June 2016

DETAILED DESCRIPTION:
BACKGROUND/INTRODUCTION:

Recently, multiple modalities of progesterone analogues have been investigated and successfully used to treat complex atypical hyperplasia (CAH) and stage 1A, grade 1 endometrial adenocarcinoma. This body of research focuses on pre-menopausal women with the primary goal of preserving fertility by delaying or avoiding surgical therapy. Across multiple case series, the average time to complete response (CR: typically defined as the absence of hyperplasia, atypia or neoplasia on a follow-up biopsy specimen) is 5-9 months with 60-70% overall complete response rate and approximately 50% durable complete response rate (defined as complete histologic response with no relapse of disease over the period of time studied). There have been no published randomized controlled trials to evaluate which modality of progesterone therapy is the most efficacious, and there is no consistent retrospective data to suggest superiority of any given progesterone analogue or method of administration.

Multiple pathologic predictors of complete response to progesterone therapy have been identified. In a recent study, Gunderson found that an interval decrease in glandular cellularity on endometrial biopsy after treatment with progesterone therapy was an independent predictor of future complete response. While both decreased mitotic index and decreased glandular cellularity were significant findings in this study, only decreased glandular cellularity was independently predictive of future complete response on multivariate analysis.

Despite this growing body of evidence supporting the safety and feasibility of progesterone analogues as medical management for CAH and early-stage endometrial adenocarcinoma, little is known about its potential role as neoadjuvant chemotherapy. A recent multicenter collaborative trial coordinated by the Gynecologic Oncology Group evaluated the effect of 400mg intramuscular medroxyprogesterone acetate administered 21-24 days prior to scheduled hysterectomy for endometrioid adenocarcinoma of the uterus. Upon comparing patients' post-hysterectomy slides to pre-treatment slides, this study found a partial histologic response rate of 63% among the 59 study subjects using pre-defined criteria modified from Wheeler 2007. A down-regulation of progesterone receptor, progesterone receptor beta, Bcl-2, and Ki-67 was also noted in post-hysterectomy specimens, with lower pre-treatment levels of Ki-67 being significantly associated with increased likelihood of histologic response. No clinical data such as patient characteristics, final tumor stage, or specific surgical procedure (ie lymphadenectomy) were collected.

The question of progesterone analogues as neoadjuvant chemotherapy is especially important given recent data showing that delayed time to surgery for endometrial cancer (defined as greater 12 weeks) was significantly associated with decreased 5-year survival rates. The same group of authors also found, alarmingly, that wait times in their province of Ontario, Canada more than doubled between 2000 and 2009. In this study, more than half of hysterectomies performed for endometrial cancer were not within the recommended limit of six weeks from diagnosis to surgery.

Considering the above data, treatment with a progesterone analogue prior to hysterectomy can be viewed as either a maintenance therapy or a temporizing measure, with the primary goal of preventing disease progression in those awaiting surgery rather than curative intent. This potential application of progesterone analogues may be particularly relevant in settings where women can expect a long wait time prior to definitive surgical management. There is empiric basis for this usage of DMPA, as one particularly intriguing study found that in vivo injection of MPA elevated the expression of a known metastasis suppressor gene in a murine breast cancer model.

Depot medroxyprogesterone acetate is a safe, well-studied and well-tolerated method of contraception that has been used globally since the 1960s. It does not require refrigeration and can be safely administered in remote settings with poor infrastructure, as demonstrated by its widespread use as contraception in the developing world. A history of using DMPA for contraception is believed by the World Health Organization to reduce the prevalence of endometrial cancer by 80%, with a protective period of at least 8 years after cessation. Apart from GOG 211, depot medroxyprogesterone acetate's role as a potential neoadjuvant chemotherapeutic agent has not been studied in isolation; rather it has been grouped with other progesterone analogues in retrospective trials of fertility-sparing agents for CAH or endometrial cancer.

Depot medroxyprogesterone acetate is used in the 150mg dose for contraception, however it has been used at higher doses of up to 1000mg weekly for several months in the setting of malignancy with no short-term side effects noted in these studies. More recently, a single dose of 400mg DMPA was compared to venlafaxine to treat women with bothersome hot flashes; at 6 weeks DMPA was superior at reducing hot flashes and associated with less short-term toxicity. GOG 211 used a one-time 400mg dose for maximal progestin effect.

DATA COLLECTION/INTERPRETATION: All data will be collected by the research assistant or study physician. The study drug will be administered during the patient's first visit at the Program in Women's Oncology after the decision is made to undergo hysterectomy for complex atypical hyperplasia or grade 1 or grade 2 endometrioid adenocarcinoma. Prior to injection with the study drug, a questionnaire will be completed by the patient to identify any factors that may influence histologic response to depot medroxyprogesterone acetate as well as baseline demographic information: age, race/ethnicity, education level, gravidity and parity, height/weight and body mass index, diabetes, hypertension, polycystic ovarian syndrome, history of irregular menses, history of oral contraceptive use, menopausal status, age at menarche, family history of uterine or ovarian malignancy, family history of colorectal cancer, smoking history, personal history of malignancy and type, history of abnormal uterine bleeding and duration, recent weight loss, recent symptoms of abdominal distension, and recent symptoms of nausea/vomiting.

FACILITIES: All patient related aspects of the study will transpire in the Women and Infants Program in Women's Oncology outpatient clinic, Women and Infants Hospital inpatient facilities, and the Women and Infants Pathology Department. Data will initially be collected at the patient's first visit with the Women and Infants Program in Women's Oncology when the decision is made to proceed with hysterectomy. Data will be collected one more time while the patient is being prepared for surgery as an inpatient at Women and Infants Hospital. Biopsy specimens and hysterectomy specimens will be reviewed by two study pathologists at the Women and Infants Hospital Department of Pathology. Data processing and interpretation will take place at Women and Infants Hospital in conjunction with the Division of Research.

CONFIDENTIALITY: The patients enrolled in the study will be asked permission for access to their medical records. To ensure patient confidentiality, all forms will be marked with only the participant ID number, with a key containing identifying information kept separately in a locked cabinet that only research personnel will have access to. Electronic data will be stored on the Care New England file server, a file server that is located in a physically secured data center. Access to Care New England data center is card-controlled and all access to the server room is recorded. Care New England computer account management policies and practices ensure that computer access to the study database will be limited to key study personnel.

SAFETY: Study personnel will meet to review safety issues and logistics at 25%, 50% and 75% recruitment. Adverse events and complications will be recorded on the data collection sheet which will be reviewed by the PI on a rolling basis. Any adverse events associated with depot medroxyprogesterone acetate use will be reported to the IRB and the FDA by the PI or co-investigators. Depot medroxyprogesterone acetate is a routinely used medication for birth control and as medical treatment for uterine fibroids and early endometrial cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patient at the Women and Infants Program in Women's Oncology
* Biopsy-proven complex atypical hyperplasia or grade 1 or grade 2 endometrial adenocarcinoma with endometrioid histology
* Disease clinically confined to the uterus (no physical exam findings or imaging to suggest extrauterine disease)
* Ages 18 and older
* Plan for hysterectomy at Women and Infants Hospital of Rhode Island
* Able to read English or Spanish
* Able to give informed consent for involvement in the study

Exclusion Criteria:

* Allergic to medroxyprogesterone acetate
* Known sensitivity to any component of depot medroxyprogesterone acetate
* History of breast cancer, hepatic disease, uncontrolled hypertension, osteoporosis or strong osteoporotic risk factors including anorexia nervosa, rheumatoid arthritis and chronic glucocorticoid use
* Treatment with any progesterone or progesterone analogue in past 12 months

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2015-02; Primary Completion 2016-03 (Actual); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Change in glandular cellularity | 2-3 weeks after hysterectomy
  Histologic analysis of glandular cellularity in hysterectomy specimens as compared to pre-hysterectomy endometrial tissue

SECONDARY OUTCOMES:
Change in mitotic index | 2-3 weeks after hysterectomy
  Histologic analysis of mitotic index in hysterectomy specimens as compared to pre-hysterectomy endometrial tissue
Histologic grade | 2-3 weeks after hysterectomy
  Histologic analysis of tumor grade in hysterectomy specimens
Depth of invasion | 2-3 weeks after hysterectomy
  Pathologic analysis of depth of invasion in hysterectomy specimens
Tumor size | 2-3 weeks after hysterectomy
  Pathologic analysis of tumor size in hysterectomy specimens
Lymph node involvement | 2-3 weeks after hysterectomy
  Pathologic analysis of lymph node involvement in surgical specimens
Lymphovascular invasion | 2-3 weeks after hysterectomy
  Pathologic analysis of lymphovascular invasion in surgical specimens
Estrogen Receptor immunohistochemistry analysis | 2-3 weeks after hysterectomy
  Immunohistochemical analysis of Estrogen Receptor status in tumor specimen
Progesterone Receptor immunohistochemistry analysis | 2-3 weeks after hysterectomy
  Immunohistochemical analysis of Progesterone Receptor status in tumor specimen
Progesterone Receptor Beta immunohistochemistry analysis | 2-3 weeks after hysterectomy
  Immunohistochemical analysis of Progesterone Receptor Beta status in tumor specimen
B-Cell-Lymphoma-2 immunohistochemistry analysis | 2-3 weeks after hysterectomy
  Immunohistochemical analysis of BCL2 status in tumor specimen
Ki-67 immunohistochemistry analysis | 2-3 weeks after hysterectomy
  Immunohistochemical analysis of Ki-67 status in tumor specimen
Caspase-3 immunohistochemistry analysis | 2-3 weeks after hysterectomy
  Immunohistochemical analysis of Casp3 status in tumor specimen
Phospho-Histone-H3 immunohistochemistry analysis | 2-3 weeks after hysterectomy
  Immunohistochemical analysis of PHH3 status in tumor specimen
Functional Assessment of Cancer Therapy - Endometrial cancer version | 1-2 hours prior to hysterectomy
  Quality of life survey FACT-En, administered 1-2 hours prior to surgery
Hemoglobin level | 12-24 hours after hysterectomy
  Hemoglobin level drawn 12-24 hours after hysterectomy to evaluate if DMPA improves blood count via diminished bleeding
Final cancer stage | 2-3 weeks after hysterectomy
  Pathologic determination of patient's definitive stage of endometrial cancer per FIGO guidelines

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Fiascone, MD, Principal Investigator — Department of medical education
Locations (1):
- Women and Infants Hospital, Program in Women's Oncology, Providence, Rhode Island, United States

REFERENCES:
- [Background] Elit LM, O'Leary EM, Pond GR, Seow HY. Impact of wait times on survival for women with uterine cancer. J Clin Oncol. 2014 Jan 1;32(1):27-33. doi: 10.1200/JCO.2013.51.3671. Epub 2013 Nov 25. PMID 24276779
- [Background] Gunderson CC, Dutta S, Fader AN, Maniar KP, Nasseri-Nik N, Bristow RE, Diaz-Montes TP, Palermo R, Kurman RJ. Pathologic features associated with resolution of complex atypical hyperplasia and grade 1 endometrial adenocarcinoma after progestin therapy. Gynecol Oncol. 2014 Jan;132(1):33-7. doi: 10.1016/j.ygyno.2013.11.033. Epub 2013 Dec 4. PMID 24316307
- [Background] Loprinzi CL, Levitt R, Barton D, Sloan JA, Dakhil SR, Nikcevich DA, Bearden JD 3rd, Mailliard JA, Tschetter LK, Fitch TR, Kugler JW. Phase III comparison of depomedroxyprogesterone acetate to venlafaxine for managing hot flashes: North Central Cancer Treatment Group Trial N99C7. J Clin Oncol. 2006 Mar 20;24(9):1409-14. doi: 10.1200/JCO.2005.04.7324. Epub 2006 Feb 27. PMID 16505409
- [Background] O'Leary E, Elit L, Pond G, Seow H. The wait time creep: changes in the surgical wait time for women with uterine cancer in Ontario, Canada, during 2000-2009. Gynecol Oncol. 2013 Oct;131(1):151-7. doi: 10.1016/j.ygyno.2013.06.036. Epub 2013 Jul 7. PMID 23838037
- [Background] Palmieri D, Halverson DO, Ouatas T, Horak CE, Salerno M, Johnson J, Figg WD, Hollingshead M, Hursting S, Berrigan D, Steinberg SM, Merino MJ, Steeg PS. Medroxyprogesterone acetate elevation of Nm23-H1 metastasis suppressor expression in hormone receptor-negative breast cancer. J Natl Cancer Inst. 2005 May 4;97(9):632-42. doi: 10.1093/jnci/dji111. PMID 15870434
- [Background] Park JY, Kim DY, Kim TJ, Kim JW, Kim JH, Kim YM, Kim YT, Bae DS, Nam JH. Hormonal therapy for women with stage IA endometrial cancer of all grades. Obstet Gynecol. 2013 Jul;122(1):7-14. doi: 10.1097/AOG.0b013e3182964ce3. PMID 23743459
- [Background] Rosenfield A, Maine D, Rochat R, Shelton J, Hatcher RA. The Food and Drug Administration and medroxyprogesterone acetate. What are the issues? JAMA. 1983 Jun 3;249(21):2922-8. PMID 6221125
- [Background] Wheeler DT, Bristow RE, Kurman RJ. Histologic alterations in endometrial hyperplasia and well-differentiated carcinoma treated with progestins. Am J Surg Pathol. 2007 Jul;31(7):988-98. doi: 10.1097/PAS.0b013e31802d68ce. PMID 17592264
- [Background] Zaino RJ, Brady WE, Todd W, Leslie K, Fischer EG, Horowitz NS, Mannel RS, Walker JL, Ivanovic M, Duska LR. Histologic effects of medroxyprogesterone acetate on endometrioid endometrial adenocarcinoma: a Gynecologic Oncology Group study. Int J Gynecol Pathol. 2014 Nov;33(6):543-53. doi: 10.1097/PGP.0000000000000177. PMID 25272292